CLINICAL TRIAL: NCT00867542
Title: Dental and Oral Findings in Israeli Children With Past IUGR - a Comprehensive Study
Brief Title: Dental and Oral Finding in Israeli Children With Past Intrauterine Growth Retardation (IUGR)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organization, Jerusalem, Israel
Other Study IDs: iugr2009HMO-CTIL
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Dental Caries
Keywords: past IUGR; ECC; oral findings in children with past IUGR
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- past IUGR: 3-4 y old children with past IUGR
  Interventions: Other: no intervention
- control: 3-4 y old healthy children
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention
  Other Names: ECC; past IUGR

SUMMARY:
oral status and early childhood caries (ecc) in israeli children with past IUGR

ELIGIBILITY:
Inclusion Criteria:

* children who were born and diagnosed with IUGR

Exclusion Criteria:

* children whos mothers have been diagnosed with diabetes or high blood pressure children with genetic disorders multiple babies pregnancy

Ages: 3 Years to 4 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 children aged 3-4 y old with IUGR in the past, 30 healthy children sex and age matched
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
oral status of children with past IUGR | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Jerusalem, Israel